CLINICAL TRIAL: NCT03192865
Title: Diaphragmatic Paralysis in Arthroscopic Shoulder Surgery: Consequences and Causes
Brief Title: Diaphragmatic Paralysis in Arthroscopic Shoulder Surgery
Status: Completed | Type: Observational
Sponsor: Clinique Medipole Garonne (Other)
Responsible Party: Principal Investigator, Dr Marty Philippe, Dr Anesthesiologist, Clinique Medipole Garonne
Other Study IDs: 2014-202
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Dyspnea; Hypoxia; Analgesia
MeSH Terms: conditions — Dyspnea; Hypoxia; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diaphragmatic paralysis/paresis group: Diaphragmatic paralysis can be associated with regional anesthesia procedure in arthroscopic shoulder surgery as phrenic nerve is close to the brachial plexus.
  Diaphragmatic paralysis will be defined using ultrasounds.
  Interventions: Procedure: diaphragmatic assessment using ultrasounds.
- No diaphragmatic paralysis/paresis group: Some strategies of peripheral nerve block are able to spare diaphragmatic paralysis.
  Interventions: Procedure: diaphragmatic assessment using ultrasounds.

INTERVENTIONS:
Procedure: diaphragmatic assessment using ultrasounds. — A diaphragmatic assessment will be performed using ultrasound. This is a pain free assessment. This assessment is commun in our unit after arthroscopic shoulder surgery.

SUMMARY:
This study aims to assess consequences and causes of hemidiaphragmatic paralysis for ambulatory arthroscopic shoulder surgery in patients with BMI ≥ 30 kg/m².

DETAILED DESCRIPTION:
This prospective observational study will screen patients with body mass index (BMI) ≥30 kg/m² undergoing acromioplasty or supraspinatus tendon repair. Occurrence of post-operative hemidiaphragmatic paralysis will be observed using M-mode ultrasonography and its consequences on patient ventilation: arterial oxygen saturation, dyspnea, success of ambulatory procedure. Causes of diaphragmatic paralysis will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All patients with body mass index ≥ 30kg/m², undergoing ambulatory arthroscopic shoulder surgery (acromioplasty and supraspinatus tendon repair) will be screened.

Exclusion Criteria:

age <18 years, brachial plexus neuropathies, severe bronchopulmonary disease, acute respiratory distress, coagulopathies, systemic glucocorticoid use, pregnancy, routine use of opioid medications, intolerance for one or more medications of the study protocol and diabetes.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with body mass index ≥ 30kg/m², undergoing ambulatory arthroscopic shoulder surgery (acromioplasty and supraspinatus tendon repair) will be screened.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2014-10-02 (Actual); Study Completion 2015-10-30 (Actual)

PRIMARY OUTCOMES:
Failure of outpatient arthroscopic shoulder surgery strategy | the first 6 hours
  failure of outpatient arthroscopic shoulder surgery strategy is communly associated with dyspnea or hypoxia due to diaphragmatic paralysis

SECONDARY OUTCOMES:
Assessment of peripheral nerve block strategy associated with diaphragmatic paralysis | the first 2 hours
  Different strategies of peripheral nerve block can be proposed for post-operative pain relief in arthroscopic shoulder surgery.
  All strategies were grouped in 3 parts:
  * Interscalene block with high volume of local anesthetics
  * Interscalene block with low volume of local anesthetics
  * distal block

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Medipole Garonne, Toulouse, France

IPD SHARING:
Plan to Share IPD: No